CLINICAL TRIAL: NCT00220935
Title: Orthotrac Pneumatic Vest: A Randomized, Controlled Trial of Treatment for Disc Herniation With Radiating Leg Pain
Brief Title: A Randomized, Controlled Trial of Treatment for Disc Herniation With Radiating Leg Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Back Institute (Other)
Collaborators: Innovative Spinal Technologies, Inc. (Industry); Orthofix Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P608
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2006-10-05 (Estimated); Status verified 2005-07

CONDITIONS: Radiating Leg Pain; Disc Protrusion
Keywords: Randomized controlled clinical trial
MeSH Terms: conditions — Intervertebral Disc Displacement

INTERVENTIONS:
Device: Orthotrac Pneumatic Vest

SUMMARY:
Hypothesis - This study is designed to evaluate the results of using the Orthotrac Pneumatic Vest versus an EZ form brace in patients with radiating leg pain from disc bulge / protrusion / herniation. Specifically, our hypothesis is that patients given the Orthotrac Pneumatic Vest (OPV) will have greater pain relief and increased self-reported functionality and fewer progressions to surgery than those using the EZ form brace.

DETAILED DESCRIPTION:
Patient Inclusion / Exclusion Criteria:

Patient's who present with low back and unilateral leg pain are potential candidates for recruitment in this study. For purposes of the research, leg pain will constitute symptoms extending down the leg beyond the knee. The contralateral side may have pain in the buttock and down the posterior thigh but not below the knee. The criteria are as follows:

Inclusion / Exclusion:

* Age 21 - 55
* Preferred no prior surgery or no spine surgery in previous 6 months.
* No neurological deficit
* VAS > 4.0
* Symptoms unresolved after 4 weeks
* Minimal antalgic lean of the trunk when initially weight bearing
* Pain aggravated by weight bearing standing / walking
* Reduced leg pain on recumbency
* MRI Confirmed disc bulge / protrusion / herniation (HNP) site consistent with symptoms - preferred.

Patient Recruitment:

A total of 150 subjects, 75 per group, are being sought for this study. The best time to capture the list of potential patients is at the inception of their diagnosis and treatment. The TBI practice is equipped with electronic scheduling, medical record and billing systems. This poses significant advantages for patient recruitment to this project. On a daily basis, the project coordinator/patient recruiters (PC/PR) can access daily schedules for new patients entering the system for all 17 TBI physicians. This can be cross-correlated later with exiting diagnosis of leg pain to ensure maximum capture of potential candidates.

Upon obtaining permission to solicit the patient, the project will be explained and signed informed consent obtained from patients who agree to participate. Non-participants will be solicited for signature to permit us to monitor their progress during the course of their treatment by administering the outcome questionnaires. Those whom do not sign consent to participate or consent to be monitored will continue with their care and be purged from the project records.

Patient Randomization and Blinding of Analysis:

At the inception of the project and prior to beginning patient recruitment, assignments for 180 participants will be blocked randomized to obtain equal numbers in each treatment group; Orthotrac (OPV) and EZ form brace (EZF). An additional 30 randomizations over the study sample size of 150 will be completed to allow for 10% drop-out rate in each group in case of patient voluntary withdrawal from participation.

Random assignments will be sealed in sequentially numbered envelopes and will be kept under lock in the office of the surgeon co-investigator . Upon patient signing of informed consent to participate, the project coordinator (PC / PR) will obtain the next consecutive sealed randomization envelope, assign the patient to the random group and deliver group assignment identification to the principal investigator (PI) for warehousing of recruitment data.

The patient will then be scheduled with the PC who will obtain appropriate demographic information and administer the outcome measures. Measures will be obtained at the same time as recruitment when ever possible. Results from the outcome measures will be sealed in an envelope, unscored, and delivered to the surgeon co-investigator for warehousing and later analysis. In order to maintain blinding of the PC / PR, she will measure the patient and fit him/her for both devices on the initial visit. The PI will have the proper device ordered according to randomization and will check fitting on its delivery.

Experimental Maneuver

Patients who qualify for this study will have persistent leg pain attributed to lumbar HNP and be under typical medical / chiropractic care. At the stage of their entry into this project, the question of surgical intervention may be a realistic alternative. The experimental maneuver will contrast the ability of the OPV vs the EZF to improve symptoms and function. Patients assigned to the OPV group will be measured by the PC / PR and fit for the device. They will receive instructions in its use QID for a minimum of 30 minutes. Patients assigned to the EZF orthotic will be fit for the device and instructed to wear it during weight bearing hours.

Patient Assessment and Outcome Measures:

At the inception of the patient into the project, either as a participant or non-participant, a baseline assessment will be performed by the PC. Reassessment will be completed at 6, 12, 26 and 52 weeks. The PC will monitor patient status and compliance with typical treatment on a weekly basis through the computerized scheduling and medical record. Telephone contact will be made on a biweekly basis to evaluate self-reported compliance with wear and determine any intervening health care service utilization or medication use using standardized phone interview methods

Assessment measures will include the following:

1. Inception baseline:

   a. Demographic b. Diagnostic c. Pre-episode work status d. Rang of Motion (ROM) i. Flexion / Extension ii. Straight leg raise e. Pain evaluation i. Pain levels (Visual analogue scale) ii. Quantitative pain drawing iii. Medication use f. Functional evaluation i. Oswestry Back Disability index ii. SF - 36
2. Follow-up evaluations:

   1. Work status
   2. Rang of Motion (ROM)

   i. Flexion / Extension ii. Straight leg raise c. Pain evaluation i. Pain levels (Visual analogue scale) ii. Quantitative pain drawing iii. Medication use d. Functional evaluation i. Oswestry Back Disability index ii. SF - 36
3. Bi-weekly telephone contacts

   1. Work status
   2. Medication use
   3. Wear compliance
   4. Other health care utilization
   5. TBI treatment sessions (PT, DC, MD, injections, surgical scheduling)

Primary outcome for this project will be quantitative pain levels, using the VAS. Monitoring of medication use is expected to support this outcome. Further primary outcome centering on functionality scores will focus on the Oswestry and SF 36. The SF36 results can be expected to be a useful adjunct in the assessment of patients with low back pain when combined with disease-specific questionnaires (3). All other measures will be used descriptively and as explanatory variables.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 - 55
* Preferred no prior surgery or no spine surgery in previous 6 months.
* VAS > 4.0
* Symptoms unresolved after 4 weeks
* Minimal antalgic lean of the trunk when initially weight bearing
* Pain aggravated by weight bearing standing / walking
* Reduced leg pain on recumbency
* MRI Confirmed disc bulge / protrusion / herniation (HNP) site consistent with symptoms - preferred.

Exclusion Criteria:

· No neurological deficit

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150
Dates: Start 2003-01; Study Completion 2006-07

PRIMARY OUTCOMES:
VAS
Oswestry
SF-36

SECONDARY OUTCOMES:
ROM
Pain drawing
Medication use
Wear compliance
Extra-protocol treatment seeking

CONTACTS AND LOCATIONS:
Overall Officials: John J. Triano, DC,PhD, Principal Investigator — Texas Back Institute
Locations (1):
- Texas Back Institute, Plano, Texas, United States